CLINICAL TRIAL: NCT02479282
Title: Effect of Natural Cesarean Section in Comparison to Traditional Cesarean Section on Maternal and Fetal Recovery
Brief Title: Effect of Natural Cesarean Section on Breastfeeding
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Samer mohamed ahmed, obstetric and gynecology resident, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: Nsc_123
Record Dates: First submitted 2015-06-13; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Natural Cesarean Section

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- group A (Other): natural cesarean section
  Interventions: Procedure: natural cesarean section
- group B (Other): traditional cesarean section
  Interventions: Procedure: traditional cesarean section

INTERVENTIONS:
Procedure: natural cesarean section
  Arms: group A
Procedure: traditional cesarean section
  Arms: group B

SUMMARY:
Effect of natural cesarean section in comparison to traditional cesarean section on maternal and fetal recovery.

ELIGIBILITY:
Inclusion Criteria:

1. primigravida or para one section
2. full term
3. cephalic
4. single baby
5. average weight
6. spinal anathesia

Exclusion Criteria:

1. High risk pregnancy.
2. Women with known or suspected fetal malformation.
3. Women with uterine malformations.
4. Breech or transverse lie.
5. Emergency caesarean section.
6. Previous two or more caesarean section

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-06; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
time to start breastfeeding | 3 hrs